CLINICAL TRIAL: NCT01692886
Title: A Phase 3, Randomized, Active-controlled Trial Evaluating the Safety, Tolerability, and Immunogenicity of a 13vPnC Vaccine Compared With a 7vPnC in Healthy Infants in China
Brief Title: A Study Evaluating 13-Valent Pneumococcal Conjugate Vaccine (13vPnC) In Healthy Infants In China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B1851015; 6096A1-3019
Record Dates: First submitted 2012-07-11; First posted 2012-09-25 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Pneumococcal Infection
Keywords: 13vPnC; 7vPnC; Healthy subjects; China
MeSH Terms: conditions — Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 7vPnC (3-, 4-, 5-, 12-Month) (Active Comparator)
  Interventions: Biological: 7-valent Pneumococcal Conjugate Vaccine
- 13vPnC (3-, 4-, 5-, 12-Month) (Experimental)
  Interventions: Biological: 13-valent Pnumococcal Conjugate vaccine
- 13vPnC (2-, 4-, 6-, 12-Month) (Experimental)
  Interventions: Biological: 13-valent Pnumococcal Conjugate vaccine
- 13vPnC (3-, 5-, 12-Month) (Experimental)
  Interventions: Biological: 13-valent Pnumococcal Conjugate vaccine

INTERVENTIONS:
Biological: 7-valent Pneumococcal Conjugate Vaccine — suspension in prefilled syringe for intramuscular injection; 0.5 mL; one dose at 3-Month Visit, 4-Month Visit, 5-Month Visit, and 12-Month Visit, respectively
  Other Names: 7vPnC
  Arms: 7vPnC (3-, 4-, 5-, 12-Month)
Biological: 13-valent Pnumococcal Conjugate vaccine — suspension in prefilled syringe for intramuscular injection; 0.5 mL; one dose at 3-Month Visit, 4-Month Visit, 5-Month Visit, and 12-Month Visit, respectively
  Other Names: 13vPnC
  Arms: 13vPnC (3-, 4-, 5-, 12-Month)
Biological: 13-valent Pnumococcal Conjugate vaccine — suspension in prefilled syringe for intramuscular injection; 0.5 mL; one dose at 2-Month Visit, 4-Month Visit, 6-Month Visit, and 12-Month Visit, respectively
  Other Names: 13vPnC
  Arms: 13vPnC (2-, 4-, 6-, 12-Month)
Biological: 13-valent Pnumococcal Conjugate vaccine — suspension in prefilled syringe for intramuscular injection; 0.5 mL; one dose at 3-Month Visit, 5-Month Visit, and 12-Month Visit, respectively
  Other Names: 13vPnC
  Arms: 13vPnC (3-, 5-, 12-Month)

SUMMARY:
This study is primarily designed to evaluate the IgG immune responses to the 13 pneumococcal serotypes induced by 13vPnC compared with the immune responses induced by 7vPnC when measured 1 month after the infant series, and to evaluate the acceptability of the safety profile of 13vPnC as measured by the incidence rates of local reactions, systemic events and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 42 to 77 days (approximately 2 months) at the time of enrollment.
2. Healthy infant as determined by medical history, physical examination, and judgment of the investigator.

Exclusion Criteria:

1. Previous vaccination with licensed or investigational pneumococcal vaccine.
2. A previous anaphylactic reaction to any vaccine or vaccine-related component.
3. Contraindication to vaccination with pneumococcal vaccines.

Ages: 42 Days to 77 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1674 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level ≥0.35 mcg/mL 1 Month After the Infant Series in Group 1 And Group 2. | 1 month after the infant series (6 Months of age)
Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level ≥0.35 mcg/mL 1 Month After the Infant Series in Group 3. | 1 month after the infant series (7 Months of age)
Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After the Infant Series in Group 1 and Group 2. | 1 month after the infant series (6 Months of age)
Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After the Infant Series in Group 3. | 1 month after the infant series (7 Months of age)
Percentage of Participants Reporting Adverse Events in Group 1 and Group 2. | Approximately 16 months from the participation into the study to the end of study
Percentage of Participants Reporting Adverse Events in Group 3 and Group 4. | Approximately 16 months from the participation into study to the end of study
Percentage of Participants Reporting Pre-Specified Local Reactions In the 7 Days After Each Pneumococcal Vaccination in Group 1 and Group 2. | Seven days after each pneumococcal vaccination dose within the period up to 12 months
Percentage of Participants Reporting Pre-Specified Local Reactions In the 7 Days After Each Pneumococcal Vaccination in Group 3 and Group 4. | Seven days after each pneumococcal vaccination dose within the period up to 12 months
Percentage of Participants Reporting Pre-Specified Systemic Events (Including The Use Of Antipyretic Medication) In the 7 Days After Each Pneumococcal Vaccination in Group 1 and Group 2. | Seven days after each pneumococcal vaccination dose within the period up to 12 months
Percentage of Participants Reporting Pre-Specified Systemic Events (Including The Use Of Antipyretic Medication) In the 7 Days After Each Pneumococcal Vaccination in Group 3 and Group 4. | Seven days after each pneumococcal vaccination dose within the period up to 12 months

SECONDARY OUTCOMES:
Percentage of Participants In A Subset Achieving Serotype-specific Opsonophagocytic Activity (OPA) Titer ≥ Lower Limit Of Quantitation (LLOQ) 1 Month After the Infant Series in Group 1 And Group 2. | 1 month after the infant series (6 Months of age)
Percentage of Participants In A Subset Achieving Serotype-specific Opsonophagocytic Activity (OPA) Titer ≥ Lower Limit Of Quantitation (LLOQ) 1 Month After the Infant Series in Group 3. | 1 month after the infant series (7 Months of age)
Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) 1 Month After the Infant Series in Group 1 and Group 2. | 1 month after the infant series (6 Months of age)
Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) 1 Month After the Infant Series in Group 3. | 1 month after the infant series (7 Months of age)
Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After the Toddler Dose in Group 2 and Group 3. | 1 month after the toddler dose (13 Months of age)
Percentage of Participants In A Subset Achieving Serotype-specific Opsonophagocytic Activity (OPA) Titer ≥ Lower Limit Of Quantitation (LLOQ) 1 Month After the Toddler Dose in Group 2 and Group 3. | 1 month after the toddler dose (13 Months of age)
Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) 1 Month After the Toddler Dose in Group 2 and Group 3. | 1 month after the toddler dose (13 Months of age)
Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level ≥0.35 mcg/mL 1 Month After the Infant Series in Group 4. | 1 month after the infant series (6 Months of age)
Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After the Infant Series in Group 4. | 1 month after the infant series (6 Months of age)
Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After the Toddler Dose in Group 4. | 1 month after the toddler dose (13 Months of age)
Percentage of Participants In A Subset Achieving Serotype-specific Opsonophagocytic Activity (OPA) Titer ≥ Lower Limit Of Quantitation (LLOQ) 1 Month After the Infant Series in Group 4. | 1 month after the infant series (6 Months of age)
Percentage of Participants In A Subset Achieving Serotype-specific Opsonophagocytic Activity (OPA) Titer ≥ Lower Limit Of Quantitation (LLOQ) 1 Month After the Toddler Dose in Group 4. | 1 month after the toddler dose (13 Months of age)
Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) 1 Month After the Infant Series in Group 4. | 1 month after the infant series (6 Months of age)
Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) 1 Month After the Toddler Dose in Group 4. | 1 month after the toddler dose (13 Months of age)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- China (4):
  - Jiangsu Province Guanyun County Center for Disease prevention and Control, Guanyun County,, Jiangsu
  - Jiangsu Province Hongze County Center for Disease prevention and Control, Huaian City, Jiangsu
  - Jiangsu Province Huaiyin District Center for Disease prevention and Control, Huaian City, Jiangsu
  - Jiangsu Province Lianshui County Center for Disease prevention and Control, Lianshui County, Jiangsu

REFERENCES:
- [Derived] Zhu F, Hu Y, Li J, Ye Q, Young MM Jr, Liang JZ, Gruber WC, Giardina PC, Scott DA. Immunogenicity and Safety of the 13-Valent Pneumococcal Conjugate Vaccine Administered in a 3 + 1 versus 2 + 1 Dose Schedule Among Infants in China. Pediatr Infect Dis J. 2019 Nov;38(11):1150-1158. doi: 10.1097/INF.0000000000002458. PMID 31626050
- [Derived] Zhu F, Hu Y, Li J, Ye Q, Young MM Jr, Zhou X, Chen Z, Yan B, Liang JZ, Gruber WC, Giardina PC, Scott DA. Immunogenicity and Safety of 13-valent Pneumococcal Conjugate Vaccine Compared With 7-valent Pneumococcal Conjugate Vaccine Among Healthy Infants in China. Pediatr Infect Dis J. 2016 Sep;35(9):999-1010. doi: 10.1097/INF.0000000000001248. PMID 27254028
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1851015&StudyName=A%20Study%20Evaluating%2013-Valent%20Pneumococcal%20Conjugate%20Vaccine%20%2813vPnC%29%20In%20Healthy%20Infants%20In%20China